CLINICAL TRIAL: NCT02514278
Title: Optimisation of Response for Organ Preservation in Rectal Cancer : Neoadjuvant Chemotherapy and Radiochemotherapy vs. Radiochemotherapy
Acronym: GRECCAR12
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2014/33
Record Dates: First submitted 2015-07-06; First posted 2015-08-03 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Rectal Cancer
Keywords: Organ preservation; Local excision; Radiochemotherapy; Neoadjuvant chemotherapy; Folfirinox; Tumour response
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy and Radiochemotherapy (Experimental): Neoadjuvant chemotherapy Folfirinox, 4 cycles:
  * oxaliplatin: 85 mg/m2
  * irinotecan: 180 mg/m²
  * folinic acid: 400 mg/m2 (DL form) or 200 mg/m2 (L form)
  * 5FU: 2400 mg/m2
  Radiochemotherapy : 2 to 4 weeks after chemotherapy, 5 weeks (50 Gy, 2 Gy/session; 25 fractions) + capecitabine (1600 mg/m2 daily 5 days/7)
  Interventions: Drug: Neoadjuvant chemotherapy Folfirinox, 4 cycles; Radiation: 50 Gy, 2 Gy/session; 25 fractions; Procedure: Local excision in good responders; Procedure: Rectal excision in bad responders; Drug: Capecitabine
- Radiochemotherapy (Active Comparator): Radiochemotherapy: 5 weeks (50 Gy, 2 Gy/session ; 25 fractions) + capecitabine (1600 mg/m2 daily 5 days/7, excluding weekends)
  Interventions: Radiation: 50 Gy, 2 Gy/session; 25 fractions; Procedure: Local excision in good responders; Procedure: Rectal excision in bad responders; Drug: Capecitabine

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy Folfirinox, 4 cycles — * oxaliplatin: 85 mg/m2
  * irinotecan: 180 mg/m²
  * folinic acid: 400 mg/m2 (DL form) or 200 mg/m2 (L form)
  * 5FU: 2400 mg/m2
  Arms: Chemotherapy and Radiochemotherapy
Radiation: 50 Gy, 2 Gy/session; 25 fractions — Radiochemotherapy 5 weeks
Procedure: Local excision in good responders — If local excision:
  * Surveillance if ypT0-1 or ypT2Nx/cN0 (no lymph node at baseline imaging)
  * Complementary rectal excision if ypT2Nx/cN1, ypT3 or R1.
Procedure: Rectal excision in bad responders
Drug: Capecitabine — 1600 mg/m2 daily 5 days/7

SUMMARY:
Standard treatment of rectal cancer is rectal excision with neoadjuvant radiochemotherapy. A new concept suggests organ preservation as an alternative to rectal excision in good responders after neoadjuvant radiochemotherapy to decrease surgical morbidity and increase quality of life. The rational is the fact that 15% of patients have sterilized tumours after radiochemotherapy for T3T4 rectal cancer. The French GRECCAR 2 trial is the first phase III trial investigating this strategy: patients with T2T3 low rectal carcinomas (size ≤4 cm) received 50 Gy with capecitabine and good clinical responders (≤2 cm) were randomized between local and rectal excision. The main findings were: the rate of complete pathologic response was higher after radiochemotherapy for small T2T3 than for T3T4 tumours (40% vs 15% ypT0) and good pathologic responders (ypT0-1) were associated with zero positive mesorectal nodes.

The objective of the new trial is to increase the proportion of patients treated with organ preservation by optimizing tumour response. As compared to Folfiri, tritherapy Folfirinox has been shown to enhance the response rate. In patients with colorectal metastases, response rate and R0 resection were twice higher, resulting in improved survival. Folfirinox also increases response and chance of R0 resection rates in initially unresectable colorectal metastases, compared to standard or intensified bi-chemotherapy regimens. Adding two months of neoadjuvant chemotherapy (Folfirinox) before radiochemotherapy, the investigators expect to increase chance of organ preservation rate, as compared to radiochemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Rectal adenocarcinoma
* cT2T3
* cN0-1 (≤ 3 positive lymph nodes or size ≤8mm)
* Tumour size ≤4 cm
* Location ≤10 cm from the anal verge
* No distant metastasis
* Patient ≥18 years
* ECOG ≤2
* Effective contraception during the study
* Patient and doctor have signed informed consent

Exclusion Criteria:

* T1 or T4
* Tumour size >4cm
* N2 (>3 positive lymph nodes or size >8mm)
* Tumour > 10 cm from the anal verge
* Distant metastasis
* Chronic intestinal inflammation and/or bowel obstruction
* Contra indication for chemotherapy and/or radiotherapy
* Previous pelvic radiotherapy or chemotherapy
* Severe renal, hepatic insufficiency (serum creatinine<30ml/min)
* Peripheral neuropathy > grade 1
* Complete or partial Dihydropyrimidine deshydrogenase (DPD) deficiency (uracilemia ≥ 16 ng/mL)
* Concomitant treatment with millepertuis, yellow fever vaccine, phenytoin or sorivudine (or chemically equivalent)
* Pregnant or breast-feeding woman.
* Persons deprived of liberty or under guardianship
* Impossibility for compliance to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of organ preservation and absence of stoma | 1 year after surgery
  Number of patients with organ preservation and absence of stoma at 1 year after surgery

SECONDARY OUTCOMES:
Compliance to treatment | From beginning of neoadjuvant treatment until surgery, expected average 20 weeks after neoadjuvant treatment
  Number of patients receiving full neoadjuvent treatment and the allocated surgery
Tolerance to treatment | From beginning of neoadjuvant treatment until 1 year after surgery
  Number of patients with adverse events
Rate of clinical complete response | At 8 weeks after neoadjuvant treatment
  To determine the rate of grade 1 : no tumor at digital examination
Rate of radiological response | At 8 weeks after neoadjuvant treatment
  To determine the rate of tumor ≤ 2 cm with TRG1-3 at MRI
Rate of complete pathologic response | At surgery, expected average 10 weeks after neoadjuvant treatment
  To determine the rate of ypT0
Correlation between radiological and clinical response | Between 8 to 10 weeks after neoadjuvant treatment
  To analyse the correlation between radiological response ( tumor ≤ 2 cm with TRG1-3 at MRI) and clinical response (grade 1)
Correlation between radiological (radiomic analysis) and pathologic response | Between 8 to 10 weeks after neoadjuvant treatment
  To analyse the correlation between radiological response ( tumor ≤ 2 cm with TRG1-3 at MRI) and pathological response (ypT0)
Rate of curative surgery | At surgery, expected average 10 weeks after neoadjuvant treatment
  To determine the rate of R0 resection
Surgical morbidity | From surgery until 1 year of follow-up
  To analyse the cumulative Clavien-Dindo at 1 year
Quality of life | From randomization until 1 year after surgery
  To examine score of questionnaires : QLQ CR-30, QLQ CR-29
Local recurrence | From surgery until 3 years of follow-up
  To determine the rate of local recurrence at 3 years
Overall survival | From surgery until 3 years of follow-up
  To determine the rate of overall survival at 3 years
Disease-free survival | From surgery until 3 years of follow-up
  To determine the rate of disease-free survival at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LAURENT, Prof., Principal Investigator — University Hospital Bordeaux, France
Locations (29):
- France (29):
  - Service de Chirurgie Digestive, CHU Amiens Picardie, Amiens
  - Service de Chirurgie Digestive, CHU de Besançon, Besançon
  - Service de Chirurgie Digestive, Hôpital Haut-Lévêque - CHU de Bordeaux, Bordeaux
  - Service de Chirurgie Digestive, Institut Bergonié, Bordeaux
  - Service de Chirurgie Digestive, CHU Estaing - CHRU Clermont Ferrand, Clermont-Ferrand
  - Service de Chirurgie Digestive, Hôpital Beaujon - APHP, Clichy
  - Service de Chirurgie Digestive, Centre Georges François Leclerc - Dijon, Dijon
  - Service de Chirurgie Digestive, Hôpital Albert Michallon - CHU de Grenoble, La Tronche
  - Service de Chirurgie Digestive, Centre Oscar Lambret - Lille, Lille
  - Service de Chirurgie Digestive, Centre Léon Bérard - Lyon, Lyon
  - Service de Chirurgie Digestive, Hôpital Lyon Sud - CHU Lyon, Lyon
  - Service de Chirurgie Digestive, CHU de la Timone - Marseille, Marseille
  - Service de Chirurgie Digestive, Institut Paoli Calmette - Marseille, Marseille
  - Service de Chirurgie Digestives, Hôpital Européen de Marseille, Marseille
  - Service de Chirurgie Digestive, Institut du Cancer de Montpellier, Montpellier
  - Service d'Oncologie et Radiothérapie, Centre Azuréen de Cancérologie, Mougins
  - Service de Chirurgie Digestive,Institut de Cancérologie de Lorraine, Nancy
  - Service de Chirurgie Digestive, Hôtel Dieu - CHU de Nantes, Nantes
  - Service de Chirurgie Digestive, CHU Carémeau - Nîmes, Nîmes
  - GH Paris Saint Joseph, Paris
  - Service de Chirurgie Digestive et Oncologique, Hôpital Bicêtre - APHP, Paris
  - Service de Chirurgie Digestive, Hôpital les Diaconnesses, Paris
  - Service de Chirurgie Digestive, Hôpital Saint-Antoine - APHP, Paris
  - Service de Chirurgie Digestive, Hôpital Saint-Louis - APHP Paris, Paris
  - Service de Chirurgie Digestive, Hôpital Pontchaillou - CHU Rennes, Rennes
  - Service de Chirurgie Digestive, Hôpital Charles Nicolle - CHU de Rouen, Rouen
  - Service de Chirurgie Digestive, Hôpital Purpan - CHU de Toulouse, Toulouse
  - Service de chirurgie digestive, CHRU de Nancy -Hôpital de Brabois, Vandœuvre-lès-Nancy
  - Département de chirurgie digestive, Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No